CLINICAL TRIAL: NCT06788132
Title: Cranberry, Hibiscus, and Vitamin C Extracts Versus Placebo in Latency of Premature Rupture of Membranes. Randomized Double-blind Clinical Trial.
Brief Title: Cranberry, Hibiscus, and Vitamin C Extracts Versus Placebo in Latency of Premature Rupture of Membranes.
Acronym: SBERRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ricardo A Gutierrez Ramirez, MD, MSc, FACOG (Other)
Collaborators: Universidad Nacional Autonoma de Honduras (Other)
Responsible Party: Sponsor-Investigator, Ricardo A Gutierrez Ramirez, MD, MSc, FACOG, Professor, Universidad Nacional Autonoma de Honduras
Organization: Universidad Nacional Autonoma de Honduras (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGO-UNAH-48-5-2025
Record Dates: First submitted 2025-01-13; First posted 2025-01-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Premature Rupture of Membranes; Fetal Complications
Keywords: Cranberry; Hibiscus; Vitamin C; Premature Rupture of membranes
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Intervention Model Description: randomized, controlled, prospective, prospective, single-center, double-blind, parallel group, efficacy and superiority clinical trial
Who Masked: Participant, Investigator
Masking Description: randomized, controlled, prospective, prospective, single-center, double-blind, parallel group, efficacy and superiority clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cranberry, hibiscus and vitamin c extracts (Experimental): 1 capsule per day will be administered, containing a combination of blueberry extract 100mg equivalent 36 mg, hibiscus extract 20 mg, vitamin C 500 mg with lactobacillus 200 MU for 10 days
  Interventions: Combination Product: Cranberry products
- Starch (Placebo Comparator): One capsule of Starch per day for 10 days
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Cranberry products — One capsule of cranberry extract 100mg equivalent 36 mg, hibiscus extract 20 mg, vitamin C 500 mg with lactobacillus 200 MU per day for 10 days
  Arms: Cranberry, hibiscus and vitamin c extracts
Other: Placebo — Starch one capsule per day for 10 days
  Arms: Starch

SUMMARY:
The main objective of this clinical trial is to evaluate the effect of cranberry, hibiscus and vitamin C extracts supplementation on the duration of the latency of premature rupture of membranes in pregnant women between 24 and 34 weeks with PROM compared to placebo administration through a randomized double-blind clinical trial, which will be carried out from July to December 2024 in the pathological hospitalization ward of the Hospital Materno Infantil, with a sample of 84 pregnant women, divided into 2 equal groups (A and B), a control group and a placebo group, where 1 capsule per day will be administered, containing a combination of blueberry extract 100mg equivalent 36 mg, hibiscus extract 20 mg, vitamin C 500 mg with lactobacillus 200 MU or a starch capsule for 10 days. In addition, routine complementary studies will be carried out and through descriptive statistics using Redcap for data tabulation and analysis, it will be possible to prove or reject the hypothesis that proposes that the use of cranberry, vitamin C and Hibiscus supplementation does not prolong the latency of premature rupture of membranes.

DETAILED DESCRIPTION:
Premature Rupture of Membranes (PROM) is the loss of the integrity of the amniotic membranes, which includes amniotic fluid leakage via the transvaginal route and manifests itself prior to the onset of labor. It has a worldwide prevalence between 2 and 4% as a complication of pregnancies, which means that it plays an important role in preterm births and maternal-fetal complications as it is a very frequent identifiable factor. Latin America is no exception, Peru has reported up to 0.31% of the total morbidities attended in the Emergency Obstetric Service. Its management can vary from expectant, pharmacological to surgical depending on factors associated with the mother and the product, for example, gestational age, clinical condition of the mother, toxic habits, among others. Epidemiological studies carried out in Mexico explain a series of factors that increase the risk of PROM. These include: maternal reproductive tract infections (bacterial vaginitis, trichomonas, gonorrhea, chlamydia and occult chorioamnioitis); behavioral factors (smoking, substance abuse, nutritional status and sexual relations); obstetric complications (multiple pregnancy, polyhydramnios, cervical incompetence, hemorrhage during pregnancy and trauma during pregnancy), as well as environmental changes (barometric pressure). On the other hand, the results of epidemiological, clinical, histological, microbiological and molecular biology studies support that focal infection and inflammation play a primary and secondary role in the pathogenesis of PROM. In 2001, the article Frequency of premature rupture of membranes in preterm labor and evaluation of short and long term management protocols in the labor and delivery room of the Honduran Institute of Social Security was published, which reported a prevalence of 20% of this condition in the study population.7% of this condition in the population studied, a situation that has improved and by 2016 the national document on Initial management and referral of obstetric and neonatal complications was adopted, which includes premature rupture of membranes and establishes a prevalence of 10% of pregnancies and 20% of cases occur in preterm gestations. PROM in preterm pregnancies is the cause of one third of preterm births and 10% of perinatal deaths; it is also associated with an increase in maternal infectious morbidity due to chorioamnionitis and puerperal infection, constituting a problem for the national health system. The present research is aimed at the interpretation and analysis of the effects observed in two groups of pregnant women diagnosed with premature rupture of membranes after the administration of cranberry extract, hibiscus and vitamin C in comparison with a group that will be administered placebo, which is consider important to know in view of the high prevalence of this pathology in our environment, since through the results new guidelines could be developed in its management that are cost effective and adapted to the availability of our institutional resources and to the condition of each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study.
* Patients who sign the informed consent form.
* Patients who can read and write.
* Patients without alterations in the cognitive system.
* Patients who had their delivery at the Maternal and Child Hospital.
* Patients with admission criteria for conservative management in the pathology ward of the Hospital Escuela.
* Patients with a single non-abnormal fetus.
* Premature rupture of membranes with pregnancy of >24.0 and <34.0 weeks of gestation.

Exclusion Criteria:

* Patients who do not wish to participate in the study
* Fetus with pulmonary anomalies, central nervous system and cardiopathies.
* Patient with chorioamnionitis.
* Premature rupture of membranes experienced within 14 days after amniocentesis or cervical cerclage placement.
* Multiple gestation.
* Delivery within 24 hours after admission.
* Intrauterine fetal death at presentation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Duration of latency | Since intervention until delivery, assessed up to 48 hours
  change in the duration of the latency of premature rupture of membranes in number of days

SECONDARY OUTCOMES:
neonatal complications | Since intervention until neonatal discharge, assessed up to 28 days.
  incidence of neonatal complications (APGAR<7 at 5 minutes, admission to neonatal ICU, respiratory distress syndrome, periventricular leukomalacia and necrotizing enterocolitis)
maternal complications | Since intervention until maternal discharge, assessed up to 30 days.
  incidence of maternal complications (puerperal fever, postpartum endometritis)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. Gutierrez Ramirez, MD, MSc., Study Director — Universidad Nacional Autonoma de Honduras
Locations (1):
- Hospital Escuela, Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: No
It is not necessary, none of the 18 HIPAA identifiers will be placed

REFERENCES:
- [Background] Gungorduk K, Asicioglu O, Gungorduk OC, Yildirim G, Besimoglu B, Ark C. Does vitamin C and vitamin E supplementation prolong the latency period before delivery following the preterm premature rupture of membranes? A randomized controlled study. Am J Perinatol. 2014 Mar;31(3):195-202. doi: 10.1055/s-0033-1343774. Epub 2013 Apr 16. PMID 23592317